CLINICAL TRIAL: NCT06987305
Title: Intravenous rhTNK-tPA Versus Placebo Before Endovascular Thrombectomy For Stroke Patient With Large Vessel Occlusion In The Extended Time Window: the BRIDGE-TNK EXTEND Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Intravenous rhTNK-tPA Before Stroke Thrombectomy in the Extended Time Window
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); China Shijiazhuang Pharmaceutical Company RECOMGEN PHARMACEUTICAL (GUANGZHOU) CO.,LTD (Unknown)
Responsible Party: Principal Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRIDGE-TNK EXTEND
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Acute Ischemic
Keywords: acute ischemic stroke; endovascular treatment; rhTNK-tPA
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhTNK-tPA group (Experimental): Patients in this group will be treated with intravenous rhTNK-tPA and endovascular thrombectomy
  Interventions: Drug: Intravenous rhTNK-tPA; Procedure: Endovascular thrombectomy
- Placebo group (Placebo Comparator): Patients in this group will be treated with intravenous placebo and endovascular thrombectomy
  Interventions: Drug: Intravenous placebo; Procedure: Endovascular thrombectomy

INTERVENTIONS:
Drug: Intravenous rhTNK-tPA — Patients will received intravenous rhTNK-tPA
  Other Names: Intravenous tenecteplase; Intravenous TNK
  Arms: rhTNK-tPA group
Drug: Intravenous placebo — Patients will received intravenous placebo
  Other Names: Intravenous placebo (a look-alike substance that contains no drug)
  Arms: Placebo group
Procedure: Endovascular thrombectomy — Patients will received endovascular thrombectomy
  Other Names: Endovascular treatment; Mechanical thrombectomy

SUMMARY:
This randomized, double-blind, placebo-controlled phase III clinical trial aims to evaluate the efficacy and safety of intravenous recombinant human tenecteplase (rhTNK-tPA) in acute ischemic stroke patients with large vessel occlusion presenting 4.5-24 hours after last known well. The study will address two primary questions: 1) Whether rhTNK-tPA enhances pre-thrombectomy reperfusion rates and improves 90-day functional outcomes compared to placebo; 2) Whether rhTNK-tPA increases the risk of symptomatic intracranial hemorrhage and mortality.

Participants will be randomized to receive either a single bolus of rhTNK-tPA (0.25 mg/kg, max 25 mg) or matching placebo administered intravenously over 5 seconds. Key assessments include repeat neuroimaging (CT/CTA or MRI/MRA) at 24 hours post-treatment to evaluate reperfusion, NIH Stroke Scale score at day 5-7, and modified Rankin Scale score assessment at 90 days. Safety monitoring will focus on hemorrhagic transformation and mortality events throughout the study period.

DETAILED DESCRIPTION:
This multicenter, phase III trial employs a randomized, double-blind, placebo-controlled design to investigate the therapeutic window extension for rhTNK-tPA in large vessel occlusion stroke. Eligible participants are adults with large vessel occlusion confirmed by vascular imaging (CTA/MRA), and salvageable brain tissue demonstrated by perfusion imaging (CTP/MRP) mismatch. Exclusion criteria include contraindications to thrombolysis, and large core infarction (>70 mL on CTP).

Patients will be randomized 1:1 to receive either weight-adjusted rhTNK-tPA (0.25 mg/kg) or placebo. All participants will undergo endovascular thrombectomy.

The primary outcome is functional independence (mRS 0-2) at 90 days. Secondary outcomes include substantial reperfusion at initial angiogram, first-pass reperfusion, final infarct volume on day 1.5 MRI/CT, etc. Safety outcomes include symptomatic intracranial hemorrhage per Heidelberg Bleeding Classification criteria within 36 hours, and 90-day mortality.

Safety monitoring includes independent adjudication of hemorrhagic events and all-cause mortality. A sample size of 820 participants provides 80% power to detect a 10% absolute difference in functional independence (α=0.05).

The trial incorporates centralized blinded outcome assessment and intention-to-treat analysis, with data oversight by an independent clinical events committee and data safety monitoring board.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Acute ischemic stroke presenting within 4.5-24 hours of last known well;
3. No significant pre-stroke functional disability: for age <80 years, pre-stroke modified Rankin scale (mRS) ≤2; for age ≥80 years, prestroke mRS ≤1;
4. Baseline NIHSS score ≥5;
5. Imaging criteria of BOTH:

   1. Occlusion on CTA/MRA in one of the following vessels: M1/M2 segment of middle cerebral artery, A1 segment of anterior cerebral artery, V4 segment of vertebral artery, basilar artery, or P1 segment of posterior cerebral artery. For A1, or P1 occlusions, vessel diameter must be ≥0.75 mm;
   2. For anterior circulation occlusion: CTP/MRP demonstrating mismatch ratio ≥1.8, absolute mismatch volume ≥15 mL, and ischemic core volume <70 mL; OR have a mismatch between the presence of an abnormal signal on MRI diffusion-weighted imaging and no visible signal change on FLAIR. For posterior circulation occlusion: pc-ASPECTS score ≥6.
6. Plan to received endovascular thrombectomy;
7. The patient or their legal representative provides written informed consent.

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by CT/MRI;
2. Already received intravenous thrombolytic after index stroke.;
3. Pregnancy or lactation;
4. Concurrent participation in other investigation drug clinical trials;
5. Arterial tortuosity or other vascular anomalies precluding endovascular access to target vessel;
6. Pre-existing neurological/psychiatric disorders interfering with neurological assessment;
7. Space-occupying intracranial tumors (except small meningiomas ≤3 cm);
8. Intracranial aneurysm or arteriovenous malformation;
9. Terminal illness with life expectancy <6 months;
10. Anticipated inability to complete follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients functionally independent (mRS score 0 to 2) at 90 days | 90 days post-randomization
  functional independence

SECONDARY OUTCOMES:
Substantial reperfusion (defined as an eTICI grade of 2b, 2c, or 3) at initial angiogram | within 5 minutes at initial angiogram
  The expanded Thrombolysis In Cerebral Infarction (eTICI) reperfusion grading system is a 6-point scale: 0 indicates no reperfusion noted; 1, reduction in thrombus without filling of distal arterial branches; 2a, reperfusion of <50% of the territory; 2b, a reperfusion of ≥50% of the territory; 2c, near-complete perfusion with distal slow flow or presence of small cortical emboli; and 3, complete reperfusion. Successful reperfusion at initial angiogram prior to thrombectomy was defined as an eTICI grade of 2b, 2c, or 3 on the first intracranial angiogram.
Successful reperfusion (defined as an eTICI grade of 2b, 2c, or 3) at end-of-procedure angiography | 15 minutes after initial angiogram
  The expanded Thrombolysis In Cerebral Infarction (eTICI) reperfusion grading system is a 6-point scale: 0 indicates no reperfusion noted; 1, reduction in thrombus without filling of distal arterial branches; 2a, reperfusion of <50% of the territory; 2b, a reperfusion of ≥50% of the territory; 2c, near-complete perfusion with distal slow flow or presence of small cortical emboli; and 3, complete reperfusion. This outcome will be evaluate at the end of procedure.
Modified first-pass reperfusion | Perioperative (After artery puncture, but the start of procedure)
  defined as Expanded Treatment in Cerebral Infarction 2b, 2c, or 3 after the first thrombectomy pass
First-pass reperfusion | Perioperative (After artery puncture, but the start of procedure)
  defined as Expanded Treatment in Cerebral Infarction 2c, or 3 after the first thrombectomy pass
Final infarct volume on day 1.5 MRI/CT | 1.5 days post-randomization
  Infarct volume quantified via MRI/CT , with manual correction by certified radiologists.
Symptomatic intracranial hemorrhage within 48 hours | within 48 hours after endovascular treatment
  evaluate intracranial hemorrhage (Heidelberg classification)
Mortality within 90 days | 90 days post-randomization
  evaluate death rate of the two treatment groups
Procedural-related complications | within 90 days
  evaluate complications
Severe adverse events | within 90 days
  evaluate any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Qingwu Yang, MD, Principal Investigator — Department of Neurology, Xinqiao Hospital of the Army Medical University; Daojun Hong, MD, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (4):
- China (4):
  - Wuhan No. 1 Hospital, Wuhan, Hubei
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: Yes
study data without patient information
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Related papers published 6 months later, the IPD will be shared
Access Criteria: yangqwmlys@l63.com

REFERENCES:
- [Background] Albers GW, Jumaa M, Purdon B, Zaidi SF, Streib C, Shuaib A, Sangha N, Kim M, Froehler MT, Schwartz NE, Clark WM, Kircher CE, Yang M, Massaro L, Lu XY, Rippon GA, Broderick JP, Butcher K, Lansberg MG, Liebeskind DS, Nouh A, Schwamm LH, Campbell BCV; TIMELESS Investigators. Tenecteplase for Stroke at 4.5 to 24 Hours with Perfusion-Imaging Selection. N Engl J Med. 2024 Feb 22;390(8):701-711. doi: 10.1056/NEJMoa2310392. Epub 2024 Feb 8. PMID 38329148
- [Background] Yogendrakumar V, Campbell BC, Churilov L, Garcia-Esperon C, Choi PM, Cordato DJ, Guha P, Sharma G, Chen C, McDonald A, Thijs V, Mamun A, Dos Santos A, Balabanski AH, Kleinig TJ, Butcher KS, Devlin MJ, O'Rourke F, Donnan GA, Davis SM, Levi CR, Ma H, Parsons MW. Extending the time window for tenecteplase by effective reperfusion of penumbral tissue in patients with large vessel occlusion: Rationale and design of a multicenter, prospective, randomized, open-label, blinded-endpoint, controlled phase 3 trial. Int J Stroke. 2025 Mar;20(3):367-372. doi: 10.1177/17474930241308660. Epub 2024 Dec 31. PMID 39654273